CLINICAL TRIAL: NCT02924402
Title: A Phase 1 Multidose Study to Evaluate the Safety and Tolerability of XmAb13676 (Plamotamab) in Patients With CD20-Expressing Hematologic Malignancies
Brief Title: Study to Evaluate Safety and Tolerability of XmAb13676 (Plamotamab) in Patients With CD20-expressing Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XmAb13676-01
Record Dates: First submitted 2016-09-14; First posted 2016-10-05 (Estimated); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: B-cell Non-Hodgkins Lymphoma; Chronic Lymphocytic Leukemia
Keywords: NHL; B-cell Prolymphocytic Leukemia; Transformed Lymphoma; Burkitt's Lymphoma; Mantle Cell Lymphoma; Hairy Cell Leukemia; Splenic Marginal Zone Lymphoma; Waldenstrom's Macroglobulinemia; Variant Hairy Cell Leukemia; Splenic B-cell Lymphoma/Leukemia; Lymphoplasmacytic Lymphoma; Extranodal Marginal Zone Lymphoma (MALT); MALT Lymphoma; Nodal Marginal Zone Lymphoma; Follicular Lymphoma; In Situ Follicular Neoplasia; Duodenal-type Follicular Lymphoma; Large B-cell Lymphoma with IRF4 rearrangement; Primary Cutaneous Follicle Center Lymphoma; Diffuse Large B-cell Lymphoma; DLBCL; T-cell/Histiocyte-Rich Large B-cell Lymphoma; Primary Cutaneous DLBCL, leg type; EBV-positive DLBCL, NOS; EBV-positive Mucocutaneous Ulcer; DLBCL Associated with Chronic Inflammation; Lymphomatoid Granulomatosis; Primary Mediastinal (Thymic) Large B-cell Lymphoma; Intravascular Large B-cell Lymphoma; ALK+ Large B-cell Lymphoma; Plasmablastic Lymphoma; Primary Effusion Lymphoma; HHV8+ DLBCL; Burkitt-like Lymphoma with 11q Aberration; High-grade B-cell Lymphoma; B-cell Lymphoma, unclassifiable; Post-transplant Lymphoproliferative Disorder; PTLD; SLL; High-grade Lymphoma; Richter's Transformation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic, B-Cell; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia; Leukemia; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Pyloric Stenosis, Hypertrophic; Lymphomatoid Granulomatosis; Plasmablastic Lymphoma; Lymphoma, Primary Effusion; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: This study will enroll two parallel disease groups in escalation: patients with non-CLL B cell malignancies and patients with CLL/SLL/Richter's Transformation. In expansion it will enroll DLBCL and FL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Non-CLL B Cell Malignancies (Group NHL) Part A (Experimental): XmAb13676 administered IV up to 8 weeks, if receiving benefit, this can be extended at investigator's discretion
  Interventions: Biological: XmAb13676
- CLL/SLL (Group CLL) Part A (Experimental): XmAb13676 administered IV up to 8 weeks, if receiving benefit, this can be extended at investigator's discretion
  Interventions: Biological: XmAb13676
- Non-CLL B Cell Malignancies (Group NHL) Part B (Experimental): XmAb13676 administered IV up to 8 weeks, if receiving benefit, this can be extended at investigator's discretion
  Interventions: Biological: XmAb13676
- CLL/SLL (Group CLL) Part B (Experimental): XmAb13676 administered IV up to 8 weeks, if receiving benefit, this can be extended at investigator's discretion
  Interventions: Biological: XmAb13676
- Non-CLL B Cell Malignancies (Group NHL) Part C / Expansion (Experimental): XmAb13676 administered IV up to 8 weeks, if receiving benefit, this can be extended at investigator's discretion
  Interventions: Biological: XmAb13676
- Non-CLL B Cell Malignancies (Group NHL) Part D / Expansion (Experimental): XmAb13676 administered SC up to 8 weeks, if receiving benefit, this can be extended at investigator's discretion
  Interventions: Biological: XmAb13676

INTERVENTIONS:
Biological: XmAb13676 — Biological

SUMMARY:
The purpose of this study is to determine the safety and tolerability of intravenous (IV) and subcutaneous (SC) administration of XmAb13676 and to determine the maximally tolerated dose (MTD) and/or recommended dose (RD).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Diagnosis of either Non-CLL B cell malignancy
* Ineligible for or have exhausted standard therapeutic options and have relapsed or refractory disease
* ECOG performance status 0-2
* Fertile patients must agree to use highly effective contraception during and for 5 months (male patients) and 8 months (female patients) after last dose of XmAb13676
* Able and willing to complete the entire study

Additional Patient Inclusion Criteria for the DLBCL Cohort (Expansion Phase)

1. Histologically confirmed diagnosis (specified by 2016 World Health Organization) of DLBCL or transformed low-grade lymphoma with measurable disease
2. Patient must be refractory or have relapsed after 2 or more standard therapeutic options, at least one of which must have included anti-CD20 antibody therapy.
3. Not a candidate for or refusing treatment with hematopoietic stem cell transplantation

Additional Patient Inclusion Criteria for the Follicular Lymphoma Cohort (Expansion Phase)

1. Diagnosis of follicular lymphoma Grades 1-3a
2. Patient must be ineligible for or have exhausted standard therapeutic options and have had 2 or more prior systemic regimens.

Exclusion Criteria:

* Cytotoxic chemotherapy, radiotherapy, or immunotherapy including other anti-CD20 antibodies within 4 weeks, or small molecule or investigational agents within 5 elimination half-lives of the first dose of XmAb13676
* Prior solid organ transplantation
* Failure to recover from Grade 3 or 4 toxicity from previous treatment
* Multiple myeloma/plasma cell leukemia or B cell acute lymphoblastic leukemia
* Known intolerance to CD20 monoclonal antibody therapy
* History of primary central nervous system lymphoma or neoplastic central nervous system disease
* Platelet count < 50 x 10^9/L
* Absolute neutrophil count < 1.0 x 10^9/L
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) at screening > 3x upper limit of normal (ULN)
* Bilirubin > 1.5 mg/dL unless prior diagnosis and documentation of ongoing hemolysis or Gilbert's syndrome has been made)
* Estimated creatinine clearance < 40 mL/min
* Active/uncontrolled autoimmune disease
* Clinically significant cardiac/cardiovascular disease, or pulmonary compromise
* Seizure disorder
* History of stroke with the past 6 mos prior to study entry
* History or evidence of a clinically unstable/uncontrollable disorder, condition or disease other than primary malignancy, that in the opinion of the Investigator would pose a risk to the patient safety or interfere with the study evaluation, procedures or completion
* Evidence of any serious bacterial, viral, parasitic or systemic fungal infections within the 30 days prior to study entry
* Positive test for human immunodeficiency virus (HIV) or hepatitis C (HCV) antibodies (unless HCV viral load test by PCR is negative)
* Positive test for HbsAg, or positive test for HBcAb (unless serology is positive due to recent intravenous immunoglobulin therapy). HBcAb positivity will be allowed if HBsAb is present or HBV-DNA is negative and patient is receiving Hep B reactivation prophylaxis.
* Patient is pregnant or breast feeding, or planning to become pregnant while enrolled in the study, and 8 months after the last dose of study drug
* Positive urine pregnancy test (ie, urine human chorionic gonadotropin) at screening
* Live viral vaccine within 2 weeks of the first dose of XmAb13676

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by the number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | Baseline Day 1 through Day 56
Identify maximum tolerated (MTD) and/or recommended dose (RD) and schedule for XmAb13676 dosing | Baseline Day 1 through Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Chet Bohac, PharmD, MD, MSc, Study Director — Executive Medical Director, Clinical Development, Xencor, Inc.
Locations (23):
- United States (10):
  - Moores UC San Diego Cancer Center, La Jolla, California
  - Mayo Clinic, Jacksonville, Florida
  - Northside Hospital, Atlanta, Georgia
  - The University of Chicago Medicine, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - The Ohio State University Wexner Medical Center and James Cancer Hospital, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - UVA Health System, Division of Hematology & Oncology, Charlottesville, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
- France (11):
  - Institut Bergonie - Centre Regional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - Hopital Henri Mondor, Créteil
  - Institut Paoli Calmette Dpt of Oncology/Hematology, Marseille
  - Chu Montpellier, Hematologie Clinique St. Eloi, Montpellier
  - CHU de Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Haut-Leveque, Service d'Hematologie Clinique et Therapie Cellulaire, Pessac
  - Centre Hospitalier Lyon-Sud, Service d'Hematologie, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CLCC Institut Gustave Roussy, Villejuif
- Gachon University Gil Medical Center, Incheon, South Korea
- Royal Marsden Hospital (RMH) - Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No